CLINICAL TRIAL: NCT02435602
Title: The Role of Narrow Band Imaging (NBI) Endoscopy Compared With Lugol Chromoendoscopy in the Early Detection of Esophageal Cancer in Patients With Prior Head and Neck Cancers: a Prospective Randomized Study
Brief Title: The Role of Chromoendoscopy in the Early Detection of Esophageal Cancer in Patients With Prior Head and Neck Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Centre of Postgraduate Medical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 506-1-09-01-14
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Esophageal Squamous Cell Carcinoma; Squamous Cell Carcinoma of the Head and Neck
Keywords: endoscopy, gastrointestinal; cancer screening
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NBI endoscopy (Active Comparator): * GI endoscopy examination and additional the entire length of esophagus is evaluate with NBI endoscopy
  * Biopsy at the visually abnormal lesions
  * Pathologic examination of all biopsy tissue specimens
  * Advises of endoscopic/surgical or oncological treatment will be given to participants who will be diagnosed with ESCC or high grade dysplasia of the esophagus.
  Interventions: Procedure: NBI endoscopy
- lugol chromoendoscopy (Active Comparator): * GI endoscopy examination and additional the entire length of esophagus is evaluate with Lugol chromoendoscopy
  * Biopsy at the unstained lesions >= 5 mm diameter
  * Pathologic examination of all biopsy tissue specimens
  * Advises of endoscopic/surgical or oncological treatment will be given to participants who will be diagnosed with ESCC or high grade dysplasia of the esophagus.
  Interventions: Procedure: Lugol chromoendoscopy

INTERVENTIONS:
Procedure: NBI endoscopy — GI endoscopy examination and additional the entire length of esophagus is evaluate with NBI endoscopy Biopsy at the visually abnormal lesions
  Arms: NBI endoscopy
Procedure: Lugol chromoendoscopy — GI endoscopy examination and additional the entire length of esophagus is evaluate with Lugol chromoendoscopy Biopsy at the unstained lesions >= 5 mm diameter Pathologic examination of all biopsy tissue specimens
  Arms: lugol chromoendoscopy

SUMMARY:
This study evaluates the role of narrow band imaging (NBI) endoscopy compared with Lugol chromoendoscopy in the early detection of esophageal cancer in patients with prior head and neck cancers.

DETAILED DESCRIPTION:
Patients with head and neck cancers have an increased risk for developing an esophageal squamous cell carcinoma (ESCC). Small, superficial, curable lesions are difficult to diagnose using only white light endoscopy. To improve detection chromoendoscopy is recommended. In this project patients are divided into two groups based on received chromoendoscopy (NBI versus Lugol). The results of two methods will be compare regarding positive predictive value to establish usage of chromoendoscopy in early detection of ESCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with past history ( >= 1 year ) of head and neck cancer treated curatively and receiving regular follow - up at the outpatient clinic of the Head and Neck Department of Maria Skłodowska - Curie Memorial Cancer Center, Institiut of Oncology
* 18 years and older
* Diagnosis of squamous cell carcinoma of oral cavity, oropharynx, hypopharynx, larynx
* Zubrod scale 0-2
* Provided written informed consent

Exclusion Criteria:

* Lack of written informed consent
* Known allergy to iodine
* Clinical conditions precluding upper GI endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Positive predictive value | 2 years
  The results of two methods are compare regarding positive predictive value.

SECONDARY OUTCOMES:
Duration of the esophagoscopy ( NBI versus Lugol staining) | 2 years
Evaluation of endoscopy ( NBI versus Lugol staining) tolerance using Visual Analogue Scale (VAS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslaw Regula, PhD, Study Director — Maria Sklodowska-Curie Memorial Cancer Center, Institiute of Oncology, Warsaw, Poland; Anna Chaber-Ciopinska, MD, Principal Investigator — Maria Sklodowska-Curie Memorial Cancer Center, Institiute of Oncology, Warsaw, Poland
Locations (1):
- Maria Sklodowska-curie Memorial Cancer Center, Institiute of Oncology, Warsaw, Poland